CLINICAL TRIAL: NCT00782821
Title: Targeted Therapy for High Immunologic Risk Renal Transplant Recipients: A Prospective, Randomized, Open-Label Pilot Study of B-Cell Depleting Therapy in Combination With Anti-Thymocyte Globulin [Rabbit] (Thymoglobulin®, Genzyme), Tacrolimus (Prograf®, Astellas), Mycophenolate Mofetil (CellCept®, Roche) and Corticosteroid Minimization
Brief Title: Randomized Trial of Induction Therapies in High Immunological Risk Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, E. Steve Woodle, MD, FACS, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: X05274
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Kidney Transplantation
Keywords: Kidney; Renal; Rejection; High risk; Induction; Immunology; Transplantation; B Cell; Allograft; Desensitization
MeSH Terms: conditions — Rejection, Psychology | interventions — thymoglobulin; Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rabbit Antithymocyte Globulin (rATG) (Active Comparator): Rabbit Antithymocyte Globulin (rATG) 1.5mg/kg per dose x 6 doses rATG was administered on post-op day 0, 2, 4, 6, 8 and 10.
  Interventions: Drug: Rabbit Antithymocyte Globulin
- RATG/Rituxan (Experimental): Rabbit Antithymocyte Globulin (rATG)/Rituxan 1.5mg/kg per dose x 5 doses of rATG. 375mg/m2 x 1 dose of rituxan. rATG was administered on post-op day 0, 2, 4, 6 and 8. Rituxan was given on post-op day 1.
  Interventions: Drug: Rabbit Antithymocyte Globulin; Drug: Rituxan
- RATG/Velcade (Experimental): Rabbit Antithymocyte Globulin (rATG) /Velcade 1.5mg/kg per dose x 5 doses of rATG. 1.3mg/m2 per dose x 4 doses of velcade. rATG was administered on post-op day 0, 2, 4, and 6. Velcade was administered on post-op day 0, 3, 7 and 10.
  Interventions: Drug: Rabbit Antithymocyte Globulin; Drug: Velcade
- RATG/Rituxan/Velcade (Experimental): Rabbit Antithymocyte Globulin (RATG) / Rituxan / Velcade 1.5mg/kg per dose x 4 doses of rATG. 200mg/m2 for 1 dose of rituxan. 1.3mg/m2 per dose x 4 doses of velcade.
  rATG was administered on post-op day 0, 2, 4, and 6. Velcade was administered on post-op day 0, 3, 7 and 10. Rituxan was given on post-op day 1.
  Interventions: Drug: Rabbit Antithymocyte Globulin; Drug: Velcade; Drug: Rituxan

INTERVENTIONS:
Drug: Rabbit Antithymocyte Globulin — rATG will be given 1.5mg/kg intravenous (IV) per dose.
  Other Names: Thymoglobulin; rATG
Drug: Velcade — Velcade will be given 1.3mg/m2 via intravenous push (IVP) per dose.
  Other Names: bortezomib
  Arms: RATG/Rituxan/Velcade; RATG/Velcade
Drug: Rituxan — Given via IV per group assignment.
  Other Names: Rituximab
  Arms: RATG/Rituxan; RATG/Rituxan/Velcade

SUMMARY:
The purpose of this research study is to find out the effects of adding B lymphocyte modulating agents in patients at risk for rejection receiving an anti-rejection (immunosuppressive) regimen of Thymoglobulin® induction with Prograf®, Cellcept® and corticosteroid therapy.

DETAILED DESCRIPTION:
Optimal induction regimens for patients at high risk for antibody and/or cell-mediated rejection have not been established. This pilot, prospective, randomized study evaluated addition of B cell/plasma cell-targeting agents to T cell-based induction with rabbit antithymocyte globulin (rATG) in high immunologic risk renal transplant recipients. Patients were randomized to induction with rATG, rATGþrituximab, rATGþbortezomib or rATGþrituximabþbortezomib.

ELIGIBILITY:
Inclusion Criteria

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Patient is between the 18 and 65 years of age, inclusive.
* Patient is considered high risk for acute rejection based on any one of the following:

  * Patient has a current Cytotoxic PRA≥ 20% or a peak Cytotoxic PRA ≥50%
  * Patient has a T or B-cell positive crossmatch (by flow cytometry) with confirmed donor-specific antibodies on solid-phase assay.
  * Historical positive serologic or cytotoxic crossmatch or DSA to donor
  * Prior allograft loss with a history of more than one acute rejection episode.
* Female subject is either postmenopausal for at least 1 year prior to initiation of study treatment, is surgically sterilized, or if of childbearing potential, agrees to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of bortezomib, or agrees to completely abstain from heterosexual intercourse. Women of childbearing potential must have a negative serum pregnancy test within the last 48 hours prior to receiving study medication.
* Male subjects, even if surgically sterilized (i.e. status post-vasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.
* Patient must have no known contraindications to treatment with bortezomib, rituximab, or thymoglobulin.

Exclusion Criteria

* Patients that have previously received or are receiving an organ transplant other than kidney.
* Patient who lost a previous allograft due to recurrence of disease
* Patient is receiving a HLA identical living related kidney transplant
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal or polyclonal antibodies
* Patients with an absolute neutrophil count of < 1,000/mm3 or platelet count < 100,000/mm3within 30 days of consent.
* Patient has Grade 2 peripheral neuropathy by CTCAE criteria within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 9.3), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any abnormality on ECG performed within 30 days of consent has to be documented by the investigator or the patient's transplant nephrologist as not medically relevant.
* Patients who are anti-HIV-positive, or HBsAg-positive or Anti-HCV positive on testing performed within one year of consent.
* Diagnosed or treated for malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Patients with current or recent severe systemic infections within the 2 weeks prior to initiation of study treatment.
* Receipt of a live vaccine within 4 weeks prior to initiation of study treatment.
* Use of other investigational drugs within 30 days or 5 half-lives prior to initiation of study treatment, whichever is longer
* Evidence of severe liver disease by medical history or physical exam with abnormal liver profile (aspartate aminotransferase [AST], alanine aminotransferase [ALT] or total bilirubin > 1.5 times upper limit of normal [ULN]) on testing performed within 30 days of consent.
* Pregnant or nursing (lactating) women and women who might become pregnant during the study. Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum -human chorionic gonadotropin pregnancy test result within the last 48 hours prior to receiving study medication. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* EBV serologic mismatch (i.e. EBV+ donor transplanted to EBV- recipient)
* CMV serologic mismatch (i.e. CMV+ donor transplanted to CMV- recipient)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Steve Woodle, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - The University Hospital, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Rabbit Antithymocyte Globulin (rATG): Thymoglobulin x 6 doses (1.5mg/kg IV).
  Thymoglobulin is to be given on post operative days (POD) 0, 2, 4, 6 in all patients. Patients who receive a 5th dose will be administered a dose of Thymoglobulin on POD 8 and those who receive a 6th dose will be administered Thymoglobulin on POD 10. All groups will receive maintenance immunosuppression consisting of tacrolimus, mycophenolate mofetil, and corticosteroids (7 day corticosteroid taper to prednisone 5 mg daily).
- RATG/Rituxan: Thymoglobulin x 5 doses (1.5mg/kg IV) + Rituximab 375mg/m2 IV
  Thymoglobulin is to be given on post operative days (POD) 0, 2, 4, 6 in all patients. Patients who receive a 5th dose will be administered a dose of Thymoglobulin on POD 8 and those who receive a 6th dose will be administered Thymoglobulin on POD 10. All groups will receive maintenance immunosuppression consisting of tacrolimus, mycophenolate mofetil, and corticosteroids (7 day corticosteroid taper to prednisone 5 mg daily).
- RATG/Velcade: Thymoglobulin x 5 doses (1.5mg/kg IV) + Velcade (1.3 mg/m2 IVP)
  Thymoglobulin is to be given on post operative days (POD) 0, 2, 4, 6 in all patients. Patients who receive a 5th dose will be administered a dose of Thymoglobulin on POD 8 and those who receive a 6th dose will be administered Thymoglobulin on POD 10. All groups will receive maintenance immunosuppression consisting of tacrolimus, mycophenolate mofetil, and corticosteroids (7 day corticosteroid taper to prednisone 5 mg daily). Patients randomized to Arm C or D will receive 1.3 mg/m2 via IVP over 3-5 minutes on POD 0, 3, 7 and 10. The dose administered on POD 0 will be administered before pre-operatively before the pre-operative dose of methylprednisolone.
- RATG/Rituxan/Velcade: Thymoglobulin x 4 doses (1.5mg/kg IV). + Rituximab 200mg/m2 IV + Bortezomib 1.3 mg/m2 IVP Thymoglobulin is to be given on post operative days (POD) 0, 2, 4, 6 in all patients. Patients who receive a 5th dose will be administered a dose of Thymoglobulin on POD 8 and those who receive a 6th dose will be administered Thymoglobulin on POD 10. All groups will receive maintenance immunosuppression consisting of tacrolimus, mycophenolate mofetil, and corticosteroids (7 day corticosteroid taper to prednisone 5 mg daily). Patients randomized to Arm C or D will receive 1.3 mg/m2 via IVP over 3-5 minutes on POD 0, 3, 7 and 10. The dose administered on POD 0 will be administered before pre-operatively before the pre-operative dose of methylprednisolone.
Period: Overall Study
Arm/Group | Rabbit Antithymocyte Globulin (rATG) | RATG/Rituxan | RATG/Velcade | RATG/Rituxan/Velcade
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 9 | 8
Not Completed | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Rabbit Antithymocyte Globulin (RATG): Thymoglobulin (RATG) x 6 doses (1.5mg/kg IV) Thymoglobulin is to be given on post operative days (POD) 0, 2, 4, 6 in all patients. Patients who receive a 5th dose will be administered a dose of Thymoglobulin on POD 8 and those who receive a 6th dose will be administered Thymoglobulin on POD 10. All groups will receive maintenance immunosuppression consisting of tacrolimus, mycophenolate mofetil, and corticosteroids (7 day corticosteroid taper to prednisone 5 mg daily).
- RATG/Rituxan: Thymoglobulin (RATG) x 5 doses (1.5mg/kg IV)+ Rituximab 375mg/m2 IV
  Thymoglobulin is to be given on post operative days (POD) 0, 2, 4, 6 in all patients. Patients who receive a 5th dose will be administered a dose of Thymoglobulin on POD 8 and those who receive a 6th dose will be administered Thymoglobulin on POD 10. All groups will receive maintenance immunosuppression consisting of tacrolimus, mycophenolate mofetil, and corticosteroids (7 day corticosteroid taper to prednisone 5 mg daily).
- RATG/Velcade: Thymoglobulin (RATG) x 5 doses (1.5mg/kg IV) + Velcade (1.3 mg/m2 IVP)
  Thymoglobulin is to be given on post operative days (POD) 0, 2, 4, 6 in all patients. Patients who receive a 5th dose will be administered a dose of Thymoglobulin on POD 8 and those who receive a 6th dose will be administered Thymoglobulin on POD 10. All groups will receive maintenance immunosuppression consisting of tacrolimus, mycophenolate mofetil, and corticosteroids (7 day corticosteroid taper to prednisone 5 mg daily).
- RATG/Rituxan/Velcade: Thymoglobulin x 4 doses (1.5mg/kg IV)+ Rituximab 200mg/m2 IV + Velcade (1.3 mg/m2 IVP)
  Thymoglobulin is to be given on post operative days (POD) 0, 2, 4, 6 in all patients. Patients who receive a 5th dose will be administered a dose of Thymoglobulin on POD 8 and those who receive a 6th dose will be administered Thymoglobulin on POD 10. All groups will receive maintenance immunosuppression consisting of tacrolimus, mycophenolate mofetil, and corticosteroids (7 day corticosteroid taper to prednisone 5 mg daily).
- Total: Total of all reporting groups
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituxan | RATG/Velcade | RATG/Rituxan/Velcade | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Full Range); unit: years] | 49.9 [46.3 to 53.8] | 52.8 [45.6 to 62.7] | 50.6 [34.5 to 63.3] | 50.1 [45.3 to 56.9] | 50.9 [34.5 to 63.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 8 | 4 | 22
  Male | 5 | 5 | 2 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40
Pre-transplant diabetes mellitus [Number; unit: participants] | 1 | 4 | 3 | 1 | 9
Dialysis pre-transplant [Number; unit: participants] | 9 | 7 | 8 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Rejection (Banff '97) or Antibody Mediated Rejection
Description: Antibody mediated rejection demonstrated to be due to, atleast in part, to anti-donor antibody at 6 months by Banff 97' criteria.
  Acute rejection IA - cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of moderate tubulitis (>4 mononuclear cells/tubular cross section or group of 10 tubular cells).
  IB - cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of severe tubulitis (>10 mononuclear cells/tubular cross section or group of 10 tubular cells) IIA - cases with mild to moderate intimal arteritis (v1) IIB - cases with server intimal arteritis comprising >25% of the luminal area (v2) III - case with transmural arteritis and/or arterial fibrinoid change and necrosis of medical smooth muscle cells (v3 with accompanying lymphoctic inflammation)
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Rabbit Antithymocyte Globulin (RATG): Thymoglobulin x 6 doses
- RATG/Rituxan: Thymoglobulin x 5 doses + Rituximab 375mg/m2
- RATG/Velcade: Thymoglobulin x 5 doses + Velcade
- RATG/Rituxan/Velcade: Thymoglobulin x 4 doses + Rituximab 200mg/m2 + Velcade
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituxan | RATG/Velcade | RATG/Rituxan/Velcade
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants | 2 | 0 | 5 | 3

2. Secondary Outcome: Antibody-mediated Rejection by Banff '97 Criteria (Updated 2005)
Description: Antibody mediated rejection demonstrated to be due to, atleast in part, to anti-donor antibody at 6 months by Banff 97' criteria. Rejection due, at least in part, to documented anti-donor antibody ('suspicious for' if antibody not demonstrated); may coincide with categories 3, 4 and 5.
  Grade I. ATN-like - C4d+, minimal inflammation Grade II. Capillary- margination and/or thromboses, C4d+ Grade III. Arterial - v3, C4d+
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituxan | RATG/Velcade | RATG/Rituxan/Velcade
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants | 1 | 0 | 3 | 1

3. Secondary Outcome: Acute Cellular Rejection by Banff '97 Criteria (Updated 2005)
Description: Acute cellular rejection IA - cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of moderate tubulitis (>4 mononuclear cells/tubular cross section or group of 10 tubular cells).
  IB - cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of severe tubulitis (>10 mononuclear cells/tubular cross section or group of 10 tubular cells) IIA - cases with mild to moderate intimal arteritis (v1) IIB - cases with server intimal arteritis comprising >25% of the luminal area (v2) III - case with transmural arteritis and/or arterial fibrinoid change and necrosis of medical smooth muscle cells (v3 with accompanying lymphoctic inflammation)
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- RATG/Velcade: Thymoglobulin x 5 doses + Bortezomib
- RATG/Rituxan/Velcade: Thymoglobulin x 4 doses + Rituximab 200mg/m2 + Bortezomib
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituxan | RATG/Velcade | RATG/Rituxan/Velcade
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants | 1 | 0 | 1 | 0

4. Secondary Outcome: Patient Survival at 12 Months
Description: Patient was still alive 12 months post study enrollment.
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Rabbit Antithymocyte Globulin (RATG): Thymoglobulin (RATG) x 6 doses (1.5mg/kg IV)
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituxan | RATG/Velcade | RATG/Rituxan/Velcade
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants | 10 | 10 | 10 | 9

5. Secondary Outcome: Patient Allograft Survival at 12 Months
Description: Patient's allograft was still functioning at 12 months post study enrollment
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Rabbit Antithymocyte Globulin (RATG): Rabbit Antithymocyte Globulin (RATG)
  Rabbit Antithymocyte Globulin (RATG): RATG
- RATG/Rituxan: Rabbit Antithymocyte Globulin (RATG)/Rituxan
  RATG/Rituxan: RATG/Rituxan
  RATG/Rituxan/Velcade: Rabbit Antithymocyte Globulin (RATG)/ Rituxan/ Velcade
- RATG/Velcade: Rabbit Antithymocyte Globulin (RATG) /Velcade
  RATG/Rituxan/Velcade: Rabbit Antithymocyte Globulin (RATG)/ Rituxan/ Velcade
- RATG/Rituxan/Velcade: Rabbit Antithymocyte Globulin (RATG) / Rituxan / Velcade
  RATG/Velcade: RATG/Velcade
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituxan | RATG/Velcade | RATG/Rituxan/Velcade
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants | 10 | 10 | 9 | 9

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituxan | RATG/Velcade | RATG/Rituxan/Velcade
Serious Adverse Events (participants affected / at risk) | 2/10 | 4/10 | 4/10 | 2/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rabbit Antithymocyte Globulin (RATG) (N=10) | RATG/Rituxan (N=10) | RATG/Velcade (N=10) | RATG/Rituxan/Velcade (N=10)
CMV +/- Status (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CMV Viremia (Infections and infestations) | 1 (1) | 3 (3) | 4 (4) | 2 (2)
CMV Invasive Disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
EBV +/- Status (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EBV Viremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EBV-related disease / PTLD (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BKV Viremia (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
BKV Nephropathy (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Other Infections (Infections and infestations) | 2 (2) | 4 (4) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rabbit Antithymocyte Globulin (RATG) (N=10) | RATG/Rituxan (N=10) | RATG/Velcade (N=10) | RATG/Rituxan/Velcade (N=10)
CTCAE Grade 1 Nausea/Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6) | 2 (2) | 3 (3)
CTCAE Grade 2 Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
CTCAE Grade 3 Nausea/Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
CTCAE Grade 1 Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 5 (5)
CTCAE Grade 2 Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3)
CTCAE Grade 3 Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes